CLINICAL TRIAL: NCT03056053
Title: Multi-center, Single-arm, Open-label Study in Patients With Insomnia Disorder to Validate the Insomnia Daytime Symptoms and Impacts Questionnaire™ (IDSIQ™)
Brief Title: Study to Validate the Questionnaire Called IDSIQ™ in Patients With Insomnia Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AC-078A203
Record Dates: First submitted 2017-01-31; First posted 2017-02-17 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Insomnia Disorder
Keywords: insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zolpidem (Other): Commercially available zolpidem (5 or 10 mg) will be administered orally once daily during the treatment period (Day 1 to Day 14) following prescribing information from each country participating in this study
  Interventions: Drug: Zolpidem

INTERVENTIONS:
Drug: Zolpidem — Commercially available tablets of zolpidem (5 or 10 mg) for oral use
  Other Names: Ambien; Zolpidem generics; Stilnox

SUMMARY:
The main study objective is to assess the content validity and the psychometric characteristics of the Insomnia Daytime Symptoms and Impacts Questionnaire™ (IDSIQ™).

DETAILED DESCRIPTION:
Zolpidem will be used as an active intervention to assess the sensitivity to change of IDSIQ™ in patients suffering from insomnia disorder.

IDSIQ™ will be administered during the screening period (within 14 days before enrollment in the study) and the treatment period (from Day 1 to Day 14). End of study (phone call) will take place 30-37 days after the end-of-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure;
* Male or female aged ≥ 18 years;
* Body mass index (BMI): 18.5 ≤ BMI (kg/m2) < 32.0;
* Insomnia disorder according to DSM-5 criteria;
* Insufficient sleep quantity evaluated according to the self-reported history and data collected in the sleep diary;
* Insomnia Severity Index score greater than or equal to 15;
* Complete the IDSIQ™ and the sleep diary questionnaire as required.

Exclusion Criteria:

* Any current history of sleep disorder other than insomnia, or any lifetime history of related breathing disorder, periodic limb movement disorder, restless legs syndrome, circadian rhythm disorder, rapid eye movement behavior disorder, or narcolepsy;
* Self-reported usual daytime napping ≥ 1 hour per day, and ≥ 3 days per week;
* Caffeine consumption ≥ 600 mg per day;
* Shift work within 2 weeks prior to the screening visit, or planned shift work from V1 to V3;
* Travel ≥ 3 time zones within 1 week prior to the screening visit, or planned travel ≥ 3 time zones from V1 to V3;
* Known severe renal impairment or know moderate or severe hepatic impairment;
* History or clinical evidence of any disease or medical condition or treatment, which may put the subject at risk of participation in the study or may interfere with the study assessments;
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Content validity of the IDSIQ™: scoring of items into domains | During the screening period, i.e. within 14 days before Day 1
  Content validity will be based on the combination of qualitative and statistical methods in order to generate a scoring algorithm

SECONDARY OUTCOMES:
Psychometric validitiy of the IDSIQ™: Internal reliability | During the screening period, i.e. within 14 days before Day 1
  Internal consistency reliability assesses the extent to which the items correlate which each other within their domain and it is evaluated by correlation scores
Psychometric validitiy of the IDSIQ™: Test-retest reliability | During the screening period, i.e. within 14 days before Day 1
  Test-retest reliability assesses the reproducibility of the domain scores during a specific time period of stable condition and it is evaluated by intraclass correlation coefficients
Psychometric validitiy of the IDSIQ™: sensitivity to change | At Week 1 and Week 2
  Changes in the IDSIQ domain scores after 2 weeks of treatment with zolpidem compared to baseline (before zolpidem administration)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Mangialaio, MD, Study Director — Actelion
Locations (9):
- United States (5):
  - Santa Monica Clinical Trials, Santa Monica, California
  - Neurotrials Research Inc, Atlanta, Georgia
  - Clinical Research CTR of Nevada, Las Vegas, Nevada
  - Clinilabs NYC, New York, New York
  - CTI Clinical Research Center, Cincinnati, Ohio
- Germany (4):
  - St-Hedwig Krankenhaus, Schlaflab, Berlin
  - Advanced Sleep Research Berlin, Berlin
  - CTC North, Universitätsklinikum Hamburg- Eppendorf, Hamburg
  - Somnibene Inst Med Forschung & Schlafmedizin, Schwerin

REFERENCES:
- [Derived] Phillips-Beyer A, Kawata AK, Kleinman L, Seboek Kinter D, Flamion B. Meaningful Within-Patient Change in Subjective Total Sleep Time in Patients with Insomnia Disorder: An Analysis of the Sleep Diary Questionnaire Using Data from Open-Label and Phase III Clinical Trials. Pharmaceut Med. 2024 Mar;38(2):133-144. doi: 10.1007/s40290-023-00512-9. Epub 2024 Feb 1. PMID 38302765
- [Derived] Hudgens S, Phillips-Beyer A, Newton L, Seboek Kinter D, Benes H. Development and Validation of the Insomnia Daytime Symptoms and Impacts Questionnaire (IDSIQ). Patient. 2021 Mar;14(2):249-268. doi: 10.1007/s40271-020-00474-z. Epub 2020 Nov 1. PMID 33131027